CLINICAL TRIAL: NCT05158205
Title: Yoga Postures and Slow, Deep Breathing in Altering Mechanistic Outcomes in Hypertension
Brief Title: Yoga in Altering Mechanistic Outcomes in Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The project period ended prior to the completion of full enrollment.
Sponsor: Texas State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7988
Record Dates: First submitted 2021-11-08; First posted 2021-12-15 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Yoga

STUDY DESIGN:
Who Masked: Participant
Masking Description: A sham control condition will be implemented if randomized to the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga postures or slow, deep breathing (Experimental)
  Interventions: Behavioral: Yoga; Behavioral: Slow, deep breathing
- Control (Sham Comparator)
  Interventions: Behavioral: Control breathing

INTERVENTIONS:
Behavioral: Yoga — 12-week yoga intervention in which 60-minute classes are completed at Texas State University 3 times per week
  Arms: Yoga postures or slow, deep breathing
Behavioral: Slow, deep breathing — 12-week home-based intervention in which 5 weekly 20-minute breathing sessions are completed
  Arms: Yoga postures or slow, deep breathing
Behavioral: Control breathing — 12-week home-based intervention in which 5 weekly 20-minute breathing sessions are completed
  Arms: Control

SUMMARY:
The proposed study will assess the effects of yoga postures and slow, deep breathing in altering oxidative stress, vascular function, and blood pressure.

DETAILED DESCRIPTION:
The purpose of this study is to determine the mechanism by which yoga lowers blood pressure in hypertensive adults.

Free radicals and enzyme activity will be analyzed from isolated immune cells and blood pressure and vascular health will be assessed at baseline and at weeks 4, 8, and 12 during the interventions or control conditions. Sedentary adults (ages 30-60 years) with elevated blood pressure or stage I hypertension will be recruited and randomized to 12 weeks of yoga, video-based breathing, or app-based breathing conditions. Yoga classes will be completed 3 times weekly at Texas State University and slow, deep breathing interventions will be completed at home 5 times weekly. Participants assigned to the app-based breathing group will also complete 5- 20-minute breathing exercises per week at home before being re-randomization at week 12. Three testing sessions will be completed at the beginning of the study: 1) familiarization and screening for elevated blood pressure or hypertension and other exclusion criteria; 2) confirmation of elevated blood pressure or hypertension via addition seated blood pressure measurements and 24-hour ambulatory blood pressure and 3-day physical activity monitoring; and 3) blood marker assessment and endothelial function measurements.

All outcomes will be measured at baseline and at 4-week intervals throughout the 12-week data collection period in all 3 groups. At each follow up visit after randomization, testing will be completed over the course of 2 sessions: 1) ambulatory blood pressure monitor and physical activity monitoring and 2) blood marker and endothelial function measurements. At the end of the waitlist sham/control period, waitlisted participants will be rerandomized to yoga or slow, deep breathing interventions. Once re-randomized, participants in each group will complete follow up testing 4,8, and 12 weeks into their respective interventions.

ELIGIBILITY:
Exclusion Criteria:

* pregnancy (tests will be administered to all premenopausal females at initial screening and follow up visits);
* having taken blood pressure or statin medications within the past 3 months (statins have been demonstrated to reduce oxidative stress);
* infection (viral or other) within the past 4 weeks;
* having adrenal or endocrine tumors (these could impact blood pressure);
* renal disease defined as an estimate glomerular filtration rate (eGFR) of less than 60 (creatinine will be tested at initial screening and eGFR will be calculated);
* hyperaldosteronism;
* prior myocardial infarction;
* known coronary heart disease;
* personal history of stroke;
* heart failure;
* cardiac arrhythmias;
* chronic obstructive pulmonary disease, asthma, or other airflow obstructions;
* recent chest pain or dyspnea;
* orthopedic limitations that preclude the execution of yoga postures;
* current insulin dependence;
* chronic inflammatory conditions (e.g., rheumatoid arthritis, lupus, HIV/AIDS, ulcerative colitis, or Crohn's disease);
* currently taking steroid or other anti-inflammatory medication;
* currently undergoing chemotherapy or radiation;
* having practiced yoga or slow, deep breathing at least once weekly within the past 6 months;
* currently smoking or having quit within the last 6 months;
* Raynaud's disease, peripheral vascular disease, or arteritis.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in peripheral blood mononuclear cell reactive oxygen species | Baseline and week 4, 8, and 12 measurements
  Blood draws will be performed at baseline and at weeks 4, 8, and 12 during the study after randomization and analyzed for free radicals after white blood cells are separated from whole blood.
Change in peripheral blood mononuclear cell NADPH oxidase cell NADPH oxidase enzyme activity | Baseline and week 4, 8, and 12 measurements
  A portion of the white blood cells isolated from a whole blood sample will be frozen and later analyzed for enzyme activity. This will be completed for blood samples obtained at baseline and weeks 4, 8, and 12.

SECONDARY OUTCOMES:
Change in 24-hour blood pressure | Baseline and week 4, 8, and 12 measurements
  An automated cuff will be worn for 24 hours while the devices takes automatic measurements every 30 minutes.
Change in flow-mediated dilation | Baseline and week 4, 8, and 12 measurements
  A cuff will placed around the forearm while an ultrasound probe is held on the upper arm to obtain a brachial artery image. The forearm cuff will be inflated for 5 minutes, then ultrasound images of the upper arm will be obtained for 3 minutes after cuff deflation.
Change in microvascular endothelial function/thermal hyperemia | Baseline and week 4, 8, and 12 measurements
  A small probe will be secured on the forearm and gradually heated for 45 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Physiology Laboratory-Texas State University, San Marcos, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided